CLINICAL TRIAL: NCT06100601
Title: Autonomic Dysfunction in Functional Dysphonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Universiteit Antwerpen (Other); University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BOF23/PDO/059
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Functional Voice Disorder; Psychogenic Voice Disorder; Muscle Tension Dysphonia
Keywords: Autonomic nervous system, functional dysphonia, heart rate variability, psychophysiology

STUDY DESIGN:
Intervention Model Description: Part 1) Case-control study Part 2) Randomized-controlled trial (3 arms)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Autonomic nervous system (ANS) regulation therapy (Experimental): HRV biofeedback is a non-invasive intervention that focuses on increasing heart rate oscillations through real-time feedback and slow-paced breathing training (Lehrer et al., 2020; Laborde et al., 2022; Pizzoli et al., 2021). Participants will practice 20 min a day (2 sessions of 10 min) for 1 month. One weekly session will be organized in the clinic under the guidance of the therapist (individual sessions), the other sessions will be organized at home, and tracked by a chest strap heart rate monitor (Polar H10) and the Elite HRV app (elitehrv.com). First, the resonance frequency (RF) (i.e. respiration rate with the highest HRV) will be personalized for each participant. Biofeedback slow-paced breathing exercises in the app will then be customized based on this RF (40% inhale, 60% exhale: e.g. 6 bpm: 4s inhale, 6s exhale). Participants will be asked to breathe in through the nose and breathe out through pursed lips, following the breath pacer with visual feedback.
  Interventions: Behavioral: ANS regulation therapy
- conventional voice therapy (CVT) (Active Comparator): The CVT will be based on Meerschman et al. (2019). This therapeutic program has been proven effective in voice therapy and is the standard clinical care for FD patients. The program is a combination of education, vocal hygiene, posture, local relaxation, costo-abdominal breathing, resonant voice, voice placing, forward focus, voice onset, semi-occluded vocal tract exercises and laryngeal manipulation. Identical to the ANS regulation therapy, participants will practice 20 min a day for 1 month. One weekly session will be organized in the clinic under the guidance of the therapist (individual sessions), the other sessions will be organized at home and tracked by the RedCap app.
  Interventions: Behavioral: conventional voice therapy (CVT)
- ANS regulation therapy + CVT (Active Comparator): The third group will receive a combination of both therapies. The same frequency and duration of practice (20 min a day for 1 month) will apply. They will also receive one weekly session in the clinic under the guidance of the therapist (individual sessions) and the other sessions will be completed at home, tracked by the Elite HRV app and the RedCap app.
  Interventions: Behavioral: ANS regulation therapy + CVT

INTERVENTIONS:
Behavioral: ANS regulation therapy — innovative intervention for functional dysphonia
  Other Names: HRV biofeedback
  Arms: Autonomic nervous system (ANS) regulation therapy
Behavioral: conventional voice therapy (CVT) — conventional voice therapy traditionally provided for functional dysphonia
  Arms: conventional voice therapy (CVT)
Behavioral: ANS regulation therapy + CVT — combination of ANS regulation therapy and CVT
  Arms: ANS regulation therapy + CVT

SUMMARY:
The first objective of this research project is to compare the occurrence and frequency of symptoms and/or disorders related to autonomic dysfunction in patients with functional dysphonia with gender- and age-matched vocally healthy controls, using a case-control study.

The second objective is to compare the effects of a novel therapy based on autonomic nervous system regulation (i.e., ANS therapy: heart rate variability biofeedback), for functional dysphonia versus coventional voice therapy (CVT) alone or in combination with ANS regulation therapy (i.e., ANS therapy + CVT), using a longitudinal randomized controlled trial (RCT).

DETAILED DESCRIPTION:
Background. Although psychological factors have been implicated in patients with functional dysphonia (FD), conventional treatment typically targets the aberrant voice symptoms exclusively. Yet, symptomatic/conventional voice therapy (CVT) is not always successful, and in view of the significant adverse quality of life (QoL) impact combined with the substantial financial burden on the healthcare system and society, research is needed to elucidate the underlying pathogenesis and psychophysiology of FD and improve treatment outcomes. Given that (1) the Vagus nerve not only innervates the larynx, but helps to regulate the autonomic nervous system (ANS), (2) autonomic dysfunction is well recognized in the fields of psychology and psychiatry, but remains relatively understudied in the area of voice disorders, and, (3) many of the psychological symptoms/features commonly observed in patients with FD may reflect ANS dysregulation, we intend to investigate ANS dysfunction as a potential psychophysiological mechanism underlying FD; and, to evaluate the comparative effectiveness of a novel therapy that aims to improve ANS regulation in patients with FD.

Objectives. The first objective of this research project is to compare the occurrence and frequency of symptoms and/or disorders related to autonomic dysfunction in patients with FD with gender- and age-matched vocally healthy controls, using a case-control study. The second objective is to compare the effects of a novel therapy based on ANS regulation (i.e., ANS therapy: heart rate variability biofeedback), for FD versus CVT alone or in combination with ANS regulation therapy (i.e., ANS therapy + CVT), using a longitudinal randomized controlled trial (RCT).

Methods. Case-control study: Autonomic (dys)function of patients with FD will be compared with gender- and age-matched vocally healthy controls, using both physiological measures (e.g. heart rate variability, skin conductance level) and psychological patient-reported outcome measures (PROMs, e.g. Neuroception of Psychological Safety Scale, Depression Anxiety and Stress Scale). RCT: The FD group will be randomly assigned to the innovative ANS therapy group, the CVT group or the ANS therapy + CVT group. All patients will receive 1 month of treatment with 20min of daily practice. Both the autonomic assessment and the voice assessment will be performed pretherapy, immediately after therapy and at 3 months follow-up by assessors blinded to group allocation and study phase.

Expected results. Higher occurrence of symptoms and/or disorders related to autonomic dysfunction are expected in patients with FD compared with vocally healthy controls. Physiological outcomes: Lower heart rate variability, lower cardiac pre-ejection period, higher respiration rate and higher skin conductance level are hypothesized in patients with FD compared with vocally healthy controls. Psychological PROMs: Higher self-report of feelings/symptoms related to autonomic dysfunction (e.g. perceived stress, anxiety) is expected in patients with FD compared with vocally healthy controls. Autonomic function is hypothesized to improve more after the ANS therapy and the ANS therapy + CVT compared with the CVT only. Voice function is expected to improve more after the ANS therapy + CVT compared with the ANS therapy and the CVT alone.

ELIGIBILITY:
Patients with functional dysphonia will be recruited from a treatment-seeking population consulting at the voice clinic of Ghent University Hospital. Inclusion criteria are all genders, all ethnicities, aged 18 - 60 years (to exclude voice-related changes due to puberty/mutation or aging/presbyphonia), diagnosed with FD by an experienced otorhinolaryngologist and SLP (defined by a voice disorder in the absence of organic or structural mucosal disease and/or neuropathology sufficient to explain the voice disturbance (Roy et al., 2003), as determined with strobovideolaryngoscopy and a multidimensional voice assessment). Exclusion criteria include: being diagnosed with an organic voice disorder, current participation in voice therapy, practice of breathing exercises including mediation and yoga, current participation in psychotherapy or physical rehabilitation, pharmacological treatment (i.e. antidepressants, antipsychotics, heart medication, antihypertensives, inhalers), previous phonosurgical interventions, lung diseases, endocrinologic diseases, metabolic diseases, cardiovascular diseases, neurologic diseases, nasal or ear diseases, pregnancy, asthma, smoking or drug consumption.

For the vocally healthy controls, inclusion criteria are all genders, all ethnicities, aged 18 - 60 years, and matched with the FD groups by age and gender. The same exclusion criteria as above apply, with the addition of: 'diagnosed with FD'.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
heart rate variability (HRV) | baseline (before the intervention), 1 months (after the intervention), 3 months follow-up
  Heart rate variability (HRV, in ms) is an autonomic index measuring the variation of the interval between consecutive heartbeats and is vagally regulated (PSA) (Thayer et al., 2009; Pizzoli et al., 2021; Singh Solorzano et al., 2022). It measures direct Vagus nerve activation potential on a cardiac level (Thayer & Lane, 2000; Sars, 2022). High HRV is associated with high vagal tone, whereas low HRV indicates ANS dysregulation with low vagal tone and SA prominence (Idrobo-Ávila et al., 2022). HRV will be determined at rest with electrocardiography using Kubios HRV analysis software (Tarvainen et al., 2002; 2014; Niskanen et al., 2004). Ag/AgCl surface electrodes will be positioned on the participant's chest in a modified lead II configuration.
Dysphonia Severity Index (DSI) | baseline (before the intervention), 1 months (after the intervention), 3 months follow-up
  The DSI is an objective multiparametric indices that quantifies voice quality (Wuyts et al., 2000)

SECONDARY OUTCOMES:
Pre-ejection period | baseline (before the intervention), 1 months (after the intervention), 3 months follow-up
  The pre-ejection period is the time between the onset of depolarization of the left ventricle and the opening of the aortic valves and will be calculated as a cardiovascular index of SA (Lozano et al., 2007)
Respiration rate | baseline (before the intervention), 1 months (after the intervention), 3 months follow-up
  Respiration rate (in bpm) will be determined via thoracic impedance (De Geus et al., 1995). For each respiratory cycle, the total cycle time between the start of inspiration and the end of expiration will be extrapolated to a per-minute respiration rate
Skin conductance level | baseline (before the intervention), 1 months (after the intervention), 3 months follow-up
  Skin conductance level (in µS) will measure the tonic electrodermal activity and reflects increased SA (Dawson et al., 2017).
The Neuroception of Psychological Safety Scale | baseline (before the intervention), 1 months (after the intervention), 3 months follow-up
  The Neuroception of Psychological Safety Scale (NPSS; Morton et al., 2022) is a psychometrically valid measure determining psychological, relational and physiological safety. It consists of 29 items subdivided into 3 subscales: compassion (e.g. I felt caring), social engagement (e.g. I felt accepted by others) and body sensations (e.g. My body felt relaxed).
The Depression Anxiety and Stress Scale 21 | baseline (before the intervention), 1 months (after the intervention), 3 months follow-up
  The Depression Anxiety and Stress Scale 21 (DASS-21; Lovibond PF & Lovibond SH, 1995; Dutch Version: De Beurs et al., 2001) is a validated 21-item checklist covering 3 subscales measuring the emotional states of depression (e.g. I felt that I had nothing to look forward to), anxiety (e.g. I felt scared with any good reason) and stress (e.g. I found myself getting agitated).
The Posttraumatic Stress Disorder Checklist for DSM-5 | baseline (before the intervention), 1 months (after the intervention), 3 months follow-up
  The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5; Weathers et al., 2013; Dutch version: Boeschoten et al., 2014; De Beurs et al., 2020) is a validated 20-item checklist that assesses the DSM-5 symptoms of PTSD. It exists of 4 clusters: re-experiencing (e.g. Repeated, disturbing dreams of the stressful experience), avoidance (e.g. Avoiding memories, thoughts, or feelings related to the stressful experience), numbing (e.g. Loss of interest in activities that you used to enjoy), and arousal factors (e.g. Irritable behavior, angry outbursts, or acting aggressively).
The short version of the Self Regulation Questionnaire | baseline (before the intervention), 1 months (after the intervention), 3 months follow-up
  The short version of the Self Regulation Questionnaire (Brown & Miller, 1999; Carey et al., 2004; Neal & Carey, 2005) is a 31-item self-report measure of the ability to self-regulate one's behavior (e.g. Once I have a goal, I can usually plan how to reach it, I have a lot of willpower).
The Pittsburgh Sleep Quality Index | baseline (before the intervention), 1 months (after the intervention), 3 months follow-up
  The Pittsburgh Sleep Quality Index (Dutch Version: Buysse et al., 1989) is a validated 19-item index assessing overall sleep quality. It consists of 7 subscales: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication and daytime dysfunction.
Laryngeal function | baseline (before the intervention), 1 months (after the intervention), 3 months follow-up
  A flexible strobovideolaryngoscopy will be performed by an experienced otorhinolaryngologist to visualize the laryngeal function and (supra)glottic activity. The video samples will be evaluated randomly and blindly by a specialized otorhinolaryngologists and SLP to assure interrater reliability; 15% of the samples will be randomly repeated to assess intrarater reliability. The Voice-Vibratory Assessment with Laryngeal Imaging (VALI) rating form (Poburka et al., 2017) will be used for these evaluations.
Acoustic Voice Quality Index (AVQI) | baseline (before the intervention), 1 months (after the intervention), 3 months follow-up
  An instrumental voice assessment will be performed by an experienced SLP, different from the therapist. Acoustic measures will be obtained by the Computerized Speech Lab (KayPENTAX, Montvale, NY) and the software program Praat (Boersma & Weenink, 2013). A Shure SM-48 and an AKG Lyra microphone will be used. Two objective multiparametric indices will quantify voice quality: the DSI (Wuyts et al., 2000) and the AVQI (Maryn et al., 2010).
Consensus Auditory Perceptual Evaluation of Voice | baseline (before the intervention), 1 months (after the intervention), 3 months follow-up
  An auditory-perceptual (subjective) voice evaluation will be performed using the Consensus Auditory Perceptual Evaluation of Voice (Kempster et al., 2009). Speech samples (sustained vowel and continuous speech) will be evaluated randomly and blindly by 2 experienced SLPs to assure interrater reliability; 15% of the samples will be randomly repeated to assess intrarater reliability.
voice-related patient-reported outcome measures | baseline (before the intervention), 1 months (after the intervention), 3 months follow-up
  The Voice Handicap Index (Jacobson et al., 1997; Dutch version: De Bodt et al., 2000), the Vocal Tract Discomfort Scale (Mathieson et al., 2009; Dutch version: Luyten et al., 2016) and the Vocal Fatigue Index (Nanjundeswaran et al., 2015) will be administered to evaluate the psychosocial impact, vocal tract discomfort and vocal fatigue associated with dysphonia.

CONTACTS AND LOCATIONS:
Overall Officials: Kristiane Van Lierde, PhD, Principal Investigator — University Ghent
Locations (1):
- Department of Rehabilitation Sciences, Ghent University (Hospital), Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No